CLINICAL TRIAL: NCT01390415
Title: A Retrospective Survey to Evaluate the Renoprotective Effect of Losartan in Type II Diabetic Patients With Microalbuminuria and Hypertension in Real Life
Brief Title: A Study to Evaluate Whether Losartan Protects the Kidney in Hypertensive Diabetic Participants With Microalbuminuria (MK0954-365 AM1)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0954-365
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Losartan 50 mg: Adults with Type II diabetes mellitus with hypertension and microalbuminuria who received losartan 50 mg for at least 6 months during the period between 1 June 2007 and 31 December 2008.
- Losartan 100 mg: Adults with Type II diabetes mellitus with hypertension and microalbuminuria who received losartan 100 mg for at least 6 months during the period between 1 June 2007 and 31 December 2008.

SUMMARY:
This study will evaluate whether losartan protects the kidney in hypertensive Type II diabetic participants with microalbuminuria.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Hypertension and has received losartan 50 mg or losartan 100 mg for at least 6 months
* Microalbuminuria (defined as microalbuminuria > 30 mg/g and < 300 mg/g by spot urine test)
* Serum creatinine ≤1.5 mg/dL for men and ≤1.4mg/dL for women
* Urinalysis with white blood cells (WBC) <5 cells per high power field
* Results of hemoglobin A1c (HbA1c), fasting blood glucose, serum creatinine, urine albumin/urine creatinine ratio and urinary analysis tests at baseline and 6 months after initiating the losartan therapy are available
* Medical history and co-morbidities (if available) listed in medical records
* Prescription information of antihypertensive regimen of losartan 50 mg or 100 mg available

Exclusion criteria:

* Treated with angiotensin-converting enzyme (ACE) inhibitors or angiotensin-receptor blockers (ARB) before initiated treatment with losartan 50 mg or losartan 100 mg
* Enrollment in another clinical trial

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with diabetes mellitus and hypertension treated with losartan 50 mg or 100 mg for at least 6 months in a hospital setting in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the medical charts of the targeted study patients were reviewed. The study index period (when patients had to have received treatment for 6 months) was from June 1st 2007 to December 31st 2008. Data were collected retrospectively.
Pre-assignment Details: 211 patients were enrolled in this study. Among these patients, 136 patients were eligible after excluding 75 patients.
Period: Overall Study
Arm/Group | Losartan 50 mg | Losartan 100 mg
Started | 99 | 37
Completed | 99 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan 50 mg | Losartan 100 mg | Total
Number analyzed (Participants) | 99 | 37 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (8.1) | 59.7 (6.0) | 59.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 16 | 55
  Male | 60 | 21 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Macroalbuminuria After 6 Months of Treatment
Description: Macroalbuminuria was defined as having an albumin/creatinine ratio (ACR) >300 mg/g and ≥30% increase from baseline.
Time Frame: Baseline and Month 6
Measure: Number; unit: participants
Arm/Group | Losartan 50 mg | Losartan 100 mg
Number analyzed (Participants) | 99 | 37
participants | 7 | 6

2. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: SBP at baseline and month 6.
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Losartan 50 mg | Losartan 100 mg
Number analyzed (Participants) | 99 | 37
mmHg
  Baseline (n=85; n=36) | 149.5 (16.0) | 145.5 (11.1)
  Month 6 (n=72; n=22) | 136.9 (14.0) | 138.4 (11.3)
  Change from Baseline at Month 6 (n=72; n=22) | -14.0 (1.6) | -7.0 (3.0)
Statistical Analysis 1: Comparison: Losartan 50 mg vs Losartan 100 mg; Between-group comparison of Change from Baseline at Month 6; Test type: Superiority or Other; p = 0.0374, t-test, 2 sided

3. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: DBP at baseline and month 6.
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Losartan 50 mg | Losartan 100 mg
Number analyzed (Participants) | 99 | 37
mmHg
  Baseline (n=85; n=36) | 85.6 (12.4) | 84.0 (8.7)
  Month 6 (n=72; n=22) | 78.2 (8.8) | 80.1 (8.2)
  Change from Baseline at Month 6 (n=72; n=22) | -9.3 (1.2) | -4.4 (2.2)
Statistical Analysis 1: Comparison: Losartan 50 mg vs Losartan 100 mg; Between-group comparison of Change from Baseline at Month 6; Test type: Superiority or Other; p = 0.0566, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Losartan 50 mg | Losartan 100 mg
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/37
Other Adverse Events (participants affected / at risk) | 0/99 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.